CLINICAL TRIAL: NCT05970770
Title: Hypotension Prediction Index Therapy is Non-inferior to Continuous Norepinephrine Infusion for Fetal Wellbeing in the Prevention of Spinal Anesthesia-Induced Hypotension for Cesarean Delivery: a Randomized Controlled Trial
Brief Title: Hypotension Prediction Index vs Norepinephrine Infusion for Prevention of Spinal Hypotension for Cesarean Delivery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPI vs NIBP
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-06

CONDITIONS: Hypotension During Surgery; Hypotension Drug-Induced
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Hypotension Prediction Index (Experimental): Patients will be monitored with Hypotension Prediction Index which will guide vasopressor therapy with boluses of norepinephrine
  Interventions: Device: Hypotension Prediction Index; Drug: Norepinephrine
- Non Invasive Blood Pressure (Active Comparator): Spinal-induced hypotension will be prevented by continuous preventive norepinephrine infusion and blood pressure will be monitored by non invasive arm cuff every minute
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Device: Hypotension Prediction Index — in addition to standard monitoring, will have hemodynamic monitoring using HemoSphere (Edwards Lifesciences, Irvine, CA; internal memory 60 gigabyte, 10 gigabyte used for operating system) with ClearSight non-invasive hemodynamic monitoring and with the Hypotension Prediction Index software enabled. They will not receive preventive vasopressors but only norepinephrine boluses if Hypotension Prediction Index >85
  Other Names: HemoSphere; Clearsight
  Arms: Hypotension Prediction Index
Drug: Norepinephrine — Patients in the HPI group will receive a norepinephrine bolus when HPI is below 85
  Other Names: noradrenaline

SUMMARY:
The goal of this randomized controlled trial is to compare for non inferiority for fetal wellbeing Hypotension Prediction Index - Guided Therapy and Continuous Norepinephrine Infusion in in the Prevention of Spinal Anesthesia-Induced Hypotension for Cesarean Delivery.

The main question it aims to answer are:

• are fetal arterial base excess comparable with the two treatments?

Participants will undergo continuous noninvasive hemodynamic monitoring with advanced Hypotension Prediction Index Researchers will compare with patients receiving continuous norepinephrine infusion and standard blood pressure monitoring with arm cuff.

DETAILED DESCRIPTION:
In the Hypotension Prediction Index group, patients will be monitored continuously with a noninvasive hemodynamic device. The Hypotension Prediction Index is a number based on al algorithm that predicts impeding hypotension if it is greater than 85. In the treatment group, patients will be treated with norepinephrine boluses if the Hypotension Prediction Index is >85. In the control group patients will be treated with preventive continuous infusion of norepinephrine and blood pressure will be measured noninvasively every minute. Data about blood pressure and the vasopressive treatment will start concomitantly to the administration of spinal anesthesia and will stop after delivery. blood gas samples will be then collected from the placental umbilical artery to compare fetal arterial base excess as primary outcome for non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the 36th and the 40th week of gestation undergoing spinal anesthesia for elective caesarian delivery.

Exclusion Criteria:

* preeclampsia;
* eclampsia;
* atrial fibrillation and sinus tachycardia;
* cardiovascular diseases;
* neuromuscular disease;
* emergent or urgent cesarean delivery;
* coagulopathies;
* contraindications to spinal anesthesia.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women at term
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Fetal Base excess | at birth
  withdrawn from umbilical fetal artery as index of perioperative metabolic acidosis

SECONDARY OUTCOMES:
Hypotensive episodes | from spinal anesthesia until delivery
  (sistolic blood pressure <80% of baseline values for <1 minute)
Total vasopressor dose | from spinal anesthesia until delivery
  total dose of micrograms administered during operation
Hypertensive episodes | from spinal anesthesia until delivery
  systolic blood pressure >140 mmHg and/or diastolic blood pressure >100 mmHg
Fetal arterial pH | at birth
  value of fetal ph at the analisys from umbilical artery withdrown at birth
Apgar score | at 5 minutes from birth
  Apgar is a quick test performed on a baby at 1 and 5 minutes after birth, examines the baby's breathing effort, heart rate, muscle tone, reflexes, skin color. Each category is scored with 0, 1, or 2, depending on the observed condition. The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano A Draisci, Prof, Principal Investigator — IRCCS fondazione policlinico universitario A. Gemelli